CLINICAL TRIAL: NCT05295719
Title: Combining Fish Oil and Exercise to Improve Obesity-associated Inflammation
Brief Title: Combining HIIT and n-3 PUFA to Reduce Inflammation and Improve Metabolic Health
Acronym: HIIT&PUFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: University of Houston (Other); Texas Tech University Health Sciences Center (Other)
Responsible Party: Principal Investigator, Kembra Albracht, Assistant Professor, Texas Tech University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-07195; GRANT12908084 (Other Grant/Funding Number: USDA NIFA)
Record Dates: First submitted 2021-12-14; First posted 2022-03-25 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Inflammation; Human Microbiome; Insulin Resistance; Dyslipidemias
MeSH Terms: conditions — Obesity; Inflammation; Insulin Resistance; Dyslipidemias | interventions — Docosahexaenoic Acids; High-Intensity Interval Training; Safflower Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo & Flexibility Training (Control) (Placebo Comparator): Subjects will take placebo (safflower oil, AlaskOmega®) for an initial supplementation period of 4 weeks. Participants will continue supplementation and will also engage in low-intensity training (control group) for 30 minutes 3 times/week for 4 weeks. All exercise sessions will be performed on a stationary bike and conducted under investigator supervision. Participants will continue supplementation and will cease low-intensity training for a 2 week follow-up period.
  Interventions: Dietary Supplement: Safflower oil; Behavioral: Low-intensity training
- Placebo & High-Intensity Interval Training (Active Comparator): Subjects will take placebo (safflower oil, AlaskOmega®) for an initial supplementation period of 4 weeks. Participants will continue supplementation and will also engage in a 4 x 4 high-intensity interval training (HIIT) exercise program 3 days/week for 4 weeks. This will include a 3 min warm up at 15% watt max followed by 4 intervals for 4 min at 65% watt max with 3 min active recovery at 15% watt max . All exercise sessions will be performed on a stationary bike and conducted under investigator supervision. Participants will continue supplementation and cease HIIT training for a 2 week follow-up period.
  Interventions: Behavioral: High-Intensity Interval Training; Dietary Supplement: Safflower oil
- n-3 PUFA & Flexibility Training (Control) (Active Comparator): Subjects will take 4 grams n-3 PUFA (AlaskOmega®) per day (3000 mg EPA and 1000 mg DHA) for an initial supplementation period of 4 weeks. Participants will continue supplementation and will also engage in low-intensity training (control group) for 30 minutes 3 times/week for 4 weeks. All exercise sessions will be performed on a stationary bike and conducted under investigator supervision. Participants will continue supplementation and cease low-intensity training for a 2 week follow-up period.
  Interventions: Dietary Supplement: Omega-3 polyunsaturated fatty acid; Behavioral: Low-intensity training
- n-3 PUFA & High-Intensity Interval Training (Experimental): Subjects will take 4 grams n-3 PUFA (AlaskOmega®) per day (3000 mg EPA and 1000 mg DHA) for an initial supplementation period of 4 weeks. Participants will continue supplementation and will also engage in a 4 x 4 high-intensity interval training (HIIT) exercise program 3 days/week for 4 weeks. This will include a 3 min warm up at 15% watt max followed by 4 intervals for 4 min at 65% watt max with 3 min active recovery at 15% watt max . All exercise sessions will be performed on a stationary bike and conducted under investigator supervision. Participants will continue supplementation and cease low-intensity training for a 2 week follow-up period.
  Interventions: Dietary Supplement: Omega-3 polyunsaturated fatty acid; Behavioral: High-Intensity Interval Training

INTERVENTIONS:
Dietary Supplement: Omega-3 polyunsaturated fatty acid — 4 grams n-3 PUFA (AlaskOmega®) per day (3000 mg EPA and 1000 mg DHA)
  Other Names: AlaskOmega
  Arms: n-3 PUFA & Flexibility Training (Control); n-3 PUFA & High-Intensity Interval Training
Behavioral: High-Intensity Interval Training — A 4 x 4 high-intensity interval training (HIIT) exercise program 3 days/week for 4 weeks. This will include a 3 min warm up at 15% watt max followed by 4 intervals for 4 min at 65% watt max with 3 min active recovery at 15% watt max.
  Other Names: HIIT
  Arms: Placebo & High-Intensity Interval Training; n-3 PUFA & High-Intensity Interval Training
Dietary Supplement: Safflower oil — 4 grams safflower oil (AlaskOmega®) per day
  Other Names: Placebo
  Arms: Placebo & Flexibility Training (Control); Placebo & High-Intensity Interval Training
Behavioral: Low-intensity training — A low-intensity training exercise program 3 days/week for 4 weeks. This will include consistently cycling at 50% HRmax for 30 min.
  Arms: Placebo & Flexibility Training (Control); n-3 PUFA & Flexibility Training (Control)

SUMMARY:
The goal of this project is to understand the combined effects of fish oil and exercise in obesity-associated inflammation. The investigators hypothesize that fish oil will improve gut bacteria profiles, which will in turn potentiate the benefits of an exercise program and improve energy utilization and reduce inflammation and metabolic risk.

DETAILED DESCRIPTION:
Incidence of obesity continues to increase in the United States and worldwide, making its prevention or reduction a public health priority. Nutrition research that can lead to effective prevention strategies is greatly needed. Inflammation is a major underlying cause for obesity, and it is imperative to understand how anti-inflammatory food sources, such as fish oil, could aid in reducing obesity. Moreover, exercise is effective at reducing systemic inflammation and improving insulin resistance. Both exercise and diet can influence health through changes in the gut microbiome; however, no studies have investigated how together these affect gut microbiome and overall metabolic health. The goal is to understand the combined effects of fish oil and exercise in obesity-associated inflammation. The investigators hypothesize that fish oil will improve gut bacteria profiles, which will in turn potentiate the benefits of an exercise program and improve energy utilization and reduce inflammation and metabolic risk. These studies will provide the foundation for development of novel strategies for obesity, inflammation, dyslipidemia and dysglycemia.

The first aim of this study will focus on determining the combined effects of n-3 PUFA and HIIT on improving metabolic risks such as obesity-related markers of inflammation, dyslipidemia, and insulin resistance.

The investigators will test the hypothesis that n-3 PUFA, in addition to HIIT, will have beneficial effects on energy utilization, as well as obesity-related markers of inflammation, dyslipidemia and insulin resistance.

Aim 2.1: Investigate the influence of n-3 PUFA and HIIT on body weight and composition Aim 2.2: Investigate the influence of n-3 PUFA and HIIT on serum markers associated with obesity Aim 2.3: Investigate influence of n-3 PUFA and HIIT on energy utilization/ markers of insulin resistance

The second aim is to determine the combined effects of n-3 polyunsaturated fatty acids (n-3 PUFA) and high-intensity interval training (HIIT) on improving gut dysbiosis.

The investigators will test the hypothesis that n-3 PUFA supplementation will improve gut microbiota composition and related metabolites, which will result in reduced inflammation and ameliorate the metabolic response to a HIIT exercise intervention in an overweight population.

Aim 1.1: Investigate the influence of n-3 PUFA and exercise on gut microbiota composition

Aim 1.2: Investigate the influence of n-3 PUFA and exercise on microbiota produced metabolites

Participants will be randomly allocated to 1 of 4 treatment groups (n = 120), each balanced for sex, BMI, lipid profile, and dietary intake. The goal is to conduct the study in smaller cohorts, such as 10-15 participants/group (n = 40-60).

Participants will first be allocated to two groups: One group will take 4 grams n-3 PUFA (AlaskOmega®) per day (3000 mg EPA and 1000 mg DHA) and one group will take placebo (safflower oil, AlaskOmega®, from Organic Technologies Inc.) for 4 weeks of initial supplementation.

Following this, one group from the treatment and one from the placebo group (creating 4 groups: (1) placebo + low-intensity training (LIT); (2) n-3 PUFA + LIT; (3) placebo + HIIT; (4) n-3 PUFA + HIIT) will also participate in a 4 x 4 HIIT exercise (4 intervals for 4 min at 85-95% HRmax with 3min active recovery at 50-70% HRmax) program utilizing cycle ergometers on 3 days/week conducted in the research lab and under investigator supervision for 4 weeks while continuing supplementation.

If not asked to exercise, participants will be instructed to maintain their normal level of physical activity but will participate in a time-matched session of low-intensity training (50% HRmax) on 3 days/week conducted in the research lab and under investigator supervision.

All participants will wear a heart rate monitor (Polar H10) provided by TTU throughout the training (HIIT and LIT) to monitor exertion level.

Capsules will be administered in a double-blind fashion and will be identical in appearance. Participants will visit the clinic to pick up capsules. To ensure compliance, subjects will be reminded via phone (text message or phone call based on participant preference) to take their capsules and counts will be conducted when they come in for study visits.

As with any acute metabolic or physiological improvements, beneficial effects of exercise on bacterial taxa and resultant metabolite production are quickly reversed with detraining. Thus, it is of interest to determine if fish consumption can ameliorate the negative metabolic and gut effects of detraining.

At the end of the 4-week intervention (week 8), participants will cease engaging in HIIT or LIT for a 2-week detraining period. Participants will continue taking their assigned supplements.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Overweight/ Obese (BMI ≥ 25 to ≤ 40 kg/m2)
* Elevated Triglycerides (>150 mg/dL)
* Prediabetes (fasting blood glucose 100 to 125 mg/dl)

Exclusion Criteria:

* Diagnosed with Diabetes or liver disease.
* Taking BP or diabetes medications.
* Received antibiotics medications in the last 6 months.
* Pregnant/ lactating/ Irregular menstrual cycle/ menopausal.
* Currently following a formal/ structured weight loss program.
* Currently taking fish oil.
* Do not have access to smart phone/ computer with internet access.
* Exercise ≥ 1 time/week or a moderate-high score on the International Physical Activity Questionnaire.
* Feeling uncomfortable riding bike for 30 minutes.
* Claustrophobic or unable to stay under the hood for metabolic testing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in Serum high-sensitivity C-reactive protein at 4 weeks | Post-Supplementation at week 4
  Serum high-sensitivity C-reactive protein (hs-CRP; mg/L)
Mean Change from Baseline in Interleukin (IL)-6 at 4 weeks | Post-Supplementation at week 4
  Interleukin (IL)-6 (pg/mL)
Mean Change from Baseline in Interleukin (IL)-10 at 4 weeks | Post-Supplementation at week 4
  Interleukin (IL)-10 (pg/mL)
Mean Change from Baseline in Monocyte chemoattractant protein-1 at 4 weeks | Post-Supplementation at week 4
  Monocyte chemoattractant protein-1 (MCP-1; pg/mL)
Mean Change from Baseline in Tumor necrosis factor at 4 weeks | Post-Supplementation at week 4
  Tumor necrosis factor (TNF)-alpha (pg/mL)
Mean Change from Baseline in Total Cholesterol at 4 weeks | Post-Supplementation at week 4
  Total cholesterol (mg/dL)
Mean Change from Baseline in High-density lipoprotein (HDL)at 4 weeks | Post-Supplementation at week 4
  High-density lipoprotein (HDL) (mg/dL)
Mean Change from Baseline in Non-high-density lipoprotein (Non-HDL) at 4 weeks | Post-Supplementation at week 4
  Non-high-density lipoprotein (Non-HDL) (mg/dL)
Mean Change from Baseline in Low-density lipoprotein (LDL) at 4 weeks | Post-Supplementation at week 4
  Low-density lipoprotein (LDL) (mg/dL)
Mean Change from Baseline in Very-low-density lipoprotein (VLDL) at 4 weeks | Post-Supplementation at week 4
  Very-low-density lipoprotein (VLDL) (mg/dL)
Mean Change from Baseline in Triglycerides at 4 weeks | Post-Supplementation at week 4
  Triglycerides (mg/dL).
Mean Change from Baseline in Total/HDL cholesterol at 4 weeks | Post-Supplementation at week 4
  Total/HDL cholesterol (mg/dL)
Mean Change from Baseline in Fasting blood glucose at 4 weeks | Post-supplementation at week 4
  Fasting blood glucose (mg/dL)
Mean Change from Baseline in Insulin at 4 weeks | Post-supplementation at week 4
  Insulin (μU/mL)
Mean Change from Baseline in Total Body Fat Percentage at 4 weeks | Post-Supplementation at week 4
  Total Body Fat Percentage (%BF): The percent of the body that is composed of fat. This will change based on the amount of fat there is as well as the amount of lean mass there is.
Mean Change from Baseline in Body Weight at 4 weeks | Post-Supplementation at week 4
  Body weight (kilograms)
Mean Change from Baseline in Skeletal Muscle Mass Percentage at 4 weeks | Post-Supplementation at week 4
  Skeletal Muscle Mass Percentage (%SMM): The percent of the body that is composed of skeletal muscle. Like %BF, this number is relative to total mass.
Mean Change from Baseline in Serum high-sensitivity C-reactive protein at 8 weeks | Post-Intervention at week 8
  Serum high-sensitivity C-reactive protein (hs-CRP; mg/L)
Mean Change from Baseline in Monocyte chemoattractant protein-1 at 8 weeks | Post-Intervention at week 8
  Monocyte chemoattractant protein-1 (MCP-1; pg/mL)
Mean Change from Baseline in Interleukin (IL)-6 at 8 weeks | Post-Intervention at week 8
  Interleukin (IL)-6 (pg/mL)
Mean Change from Baseline in Interleukin (IL)-10 at 8 weeks | Post-Intervention at week 8
  Interleukin (IL)-10 (pg/mL)
Mean Change from Baseline in Tumor necrosis factor (TNF) at 8 weeks | Post-Intervention at week 8
  Tumor necrosis factor (TNF)-alpha (pg/mL)
Mean Change from Baseline in Total Cholesterol at 8 weeks | Post-Intervention at week 8
  Total Cholesterol (mg/dL)
Mean Change from Baseline in High-density lipoprotein (HDL) at 8 weeks | Post-Intervention at week 8
  High-density lipoprotein (HDL) (mg/dL)
Mean Change from Baseline in Non-high-density lipoprotein (Non-HDL) at 8 weeks | Post-intervention at week 8
  Non-high-density lipoprotein (Non-HDL) (mg/dL)
Mean Change from Baseline in Low-density lipoprotein (LDL) at 8 weeks | Post-Intervention at week 8
  Low-density lipoprotein (LDL) (mg/dL)
Mean Change from Baseline in Very-low-density lipoprotein (VLDL) at 8 weeks | Post-Intervention at week 8
  Very-low-density lipoprotein (VLDL) (mg/dL)
Mean Change from Baseline in Triglycerides at 8 weeks | Post-Intervention at week 8
  Triglycerides (mg/dL).
Mean Change from Baseline in total/HDL cholesterol at 8 weeks | Post-Intervention at week 8
  Total/HDL cholesterol (mg/dL)
Mean Change from Baseline in Fasting blood glucose at 8 weeks | Post-Intervention at week 8
  Fasting blood glucose (mg/dL)
Mean Change from Baseline in Oral glucose tolerance test (OGTT) at 8 weeks | Post-Intervention at week 8
  Oral glucose tolerance test (OGTT). Following ingestion of 75 g oral glucose, blood samples will be drawn every 5-10 minutes for the first 30 minutes then every 30 minutes for the next 90 minutes.
Mean Change from Baseline in Insulin at 8 weeks | Post-Intervention at week 8
  Insulin (μU/mL)
Mean Change from Baseline in Body Weight at 8 weeks | Post-Intervention at week 8
  Body weight (kilograms)
Mean Change from Baseline in Total Body Fat Percentage at 8 weeks | Post-Intervention at week 8
  Total Body Fat Percentage (%BF): The percent of the body that is composed of fat. This will change based on the amount of fat there is as well as the amount of lean mass there is.
Mean Change from Baseline in Skeletal Muscle Mass Percentage at 8 weeks | Post-Intervention at week 8
  Skeletal Muscle Mass Percentage (%SMM): The percent of the body that is composed of skeletal muscle. Like %BF, this number is relative to total mass.
Mean Change from Baseline in Serum high-sensitivity C-reactive protein at 10 weeks | Post-Detraining at week 10
  Serum high-sensitivity C-reactive protein (hs-CRP; mg/L)
Mean Change from Baseline in Interleukin (IL)-6 at 10 weeks | Post-Detraining at week 10
  Interleukin (IL)-6 (pg/mL)
Mean Change from Baseline in Interleukin (IL)-10 at 10 weeks | Post-Detraining at week 10
  Interleukin (IL)-10 (pg/mL)
Mean Change from Baseline in Tumor necrosis factor (TNF) at 10 weeks | Post-Detraining at week 10
  Tumor necrosis factor (TNF)-alpha (pg/mL)
Mean Change from Baseline in Monocyte chemoattractant protein-1 at 10 weeks | Post-Detraining at week 10
  Monocyte chemoattractant protein-1 (MCP-1; pg/mL)
Mean Change from Baseline in Total Cholesterol at 10 weeks | Post-Detraining at week 10
  Total Cholesterol (mg/dL)
Mean Change from Baseline in High-density lipoprotein (HDL) at 10 weeks | Post-Detraining at week 10
  High-density lipoprotein (HDL) (mg/dL)
Mean Change from Baseline in Non-high-density lipoprotein (Non-HDL) at 10 weeks | Post-Detraining at week 10
  Non-high-density lipoprotein (Non-HDL) (mg/dL)
Mean Change from Baseline in Low-density lipoprotein (LDL) at 10 weeks | Post-Detraining at week 10
  Low-density lipoprotein (LDL)(mg/dL)
Mean Change from Baseline in Very-low-density lipoprotein (VLDL) at 10 weeks | Post-Detraining at week 10
  Very-low-density lipoprotein (VLDL) (mg/dL)
Mean Change from Baseline in Total/HDL cholesterol at 10 weeks | Post-Detraining at week 10
  Total/HDL cholesterol (mg/dL)
Mean Change from Baseline in Triglycerides at 10 weeks | Post-Detraining at week 10
  Triglycerides (mg/dL)
Mean Change from Baseline in Insulin at 10 weeks | Post-Detraining at week 10
  Insulin (μU/mL)
Mean Change from Baseline in Fasting blood glucose at 10 weeks | Post-Detraining at week 10
  Fasting blood glucose (mg/dL)
Mean Change from Baseline in Skeletal Muscle Mass Percentage at 10 weeks | Post-Detraining at week 10
  Skeletal Muscle Mass Percentage (%SMM): The percent of the body that is composed of skeletal muscle. Like %BF, this number is relative to total mass.
Mean Change from Baseline in Body weight at 10 weeks | Post-Detraining at week 10
  Body weight (kilograms)
Mean Change from Baseline in Total Body Fat Percentage at 10 weeks | Post-Detraining at week 10
  Total Body Fat Percentage (%BF): The percent of the body that is composed of fat. This will change based on the amount of fat there is as well as the amount of lean mass there is.
Mean Change from Post-Supplementation in Serum high-sensitivity C-reactive protein at 8 weeks | Post-Intervention at week 8
  Serum high-sensitivity C-reactive protein (hs-CRP; mg/L)
Mean Change from Post-Supplementation in Interleukin (IL)-6 at 8 weeks | Post-Intervention at week 8
  Interleukin (IL)-6 (pg/mL)
Mean Change from Post-Supplementation in Interleukin (IL)-10 at 8 weeks | Post-Intervention at week 8
  Interleukin (IL)-10 (pg/mL)
Mean Change from Post-Supplementation in Monocyte chemoattractant protein-1 at 8 weeks | Post-Intervention at week 8
  Monocyte chemoattractant protein-1 (MCP-1; pg/mL)
Mean Change from Post-Supplementation in Tumor necrosis factor (TNF) at 8 weeks | Post-Intervention at week 8
  Tumor necrosis factor (TNF)-alpha (pg/mL)
Mean Change from Post-Supplementation in Total Cholesterol at 8 weeks | Post-Intervention at week 8
  Total Cholesterol (mg/dL)
Mean Change from Post-Supplementation in Total/HDL cholesterol at 8 weeks | Post-Intervention at week 8
  Total/HDL cholesterol (mg/dL)
Mean Change from Post-Supplementation in High-density lipoprotein (HDL) at 8 weeks | Post-Intervention at week 8
  High-density lipoprotein (HDL) (mg/dL)
Mean Change from Post-Supplementation in Non-high-density lipoprotein (Non-HDL) at 8 weeks | Post-Intervention at week 8
  Non-high-density lipoprotein (Non-HDL) (mg/dL)
Mean Change from Post-Supplementation in Low-density lipoprotein (LDL) at 8 weeks | Post-Intervention at week 8
  Low-density lipoprotein (LDL) (mg/dL)
Mean Change from Post-Supplementation in Very-low-density lipoprotein (VLDL) at 8 weeks | Post-Intervention at week 8
  Very-low-density lipoprotein (VLDL) (mg/dL)
Mean Change from Post-Supplementation in Triglycerides at 8 weeks | Post-Intervention at week 8
  Triglycerides (mg/dL)
Mean Change from Post-Supplementation in Insulin at 8 weeks | Post-Intervention at week 8
  Insulin (μU/mL)
Mean Change from Post-Supplementation in Fasting blood glucose at 8 weeks | Post-Intervention at week 8
  Fasting blood glucose (mg/dL)
Mean Change from Post-Supplementation in Body weight at 8 weeks | Post-Intervention at week 8
  Body weight (kilograms)
Mean Change from Post-Supplementation in Total Body Fat Percentage at 8 weeks | Post-Intervention at week 8
  Total Body Fat Percentage (%BF): The percent of the body that is composed of fat. This will change based on the amount of fat there is as well as the amount of lean mass there is.
Mean Change from Post-Intervention in Serum high-sensitivity C-reactive protein at 10 weeks | Post-Detraining at week 10
  Serum high-sensitivity C-reactive protein (hs-CRP; mg/L)
Mean Change from Post-Intervention in Tumor Necrosis Factor (TNF) at 10 weeks | Post-Detraining at week 10
  Tumor necrosis factor (TNF)-alpha (pg/mL)
Mean Change from Post-Intervention in Interleukin (IL)-6 at 10 weeks | Post-Detraining at week 10
  Interleukin (IL)-6 (pg/mL)
Mean Change from Post-Intervention in Interleukin (IL)-10 at 10 weeks | Post-Detraining at week 10
  Interleukin (IL)-10 (pg/mL)
Mean Change from Post-Intervention in Monocyte Chemoattractant Protein-1 at 10 weeks | Post-Detraining at week 10
  Monocyte chemoattractant protein-1 (MCP-1; pg/mL)
Mean Change from Post-Intervention in Total Cholesterol at 10 weeks | Post-Detraining at week 10
  Total Cholesterol (mg/dL)
Mean Change from Post-Intervention in High-density lipoprotein (HDL) at 10 weeks | Post-Detraining at week 10
  High-density lipoprotein (HDL) (mg/dL)
Mean Change from Post-Intervention in Non-high-density lipoprotein (Non-HDL) at 10 weeks | Post-Detraining at week 10
  Non-high-density lipoprotein (Non-HDL) (mg/dL)
Mean Change from Post-Intervention in Low-density lipoprotein (LDL) at 10 weeks | Post-Detraining at week 10
  Low-density lipoprotein (LDL) (mg/dL)
Mean Change from Post-Intervention in Very-low-density lipoprotein (VLDL) at 10 weeks | Post-Detraining at week 10
  Very-low-density lipoprotein (VLDL) (mg/dL)
Mean Change from Post-Intervention in Total/HDL cholesterol at 10 weeks | Post-Detraining at week 10
  Total/HDL cholesterol (mg/dL)
Mean Change from Post-Intervention in Triglycerides at 10 weeks | Post-Detraining at week 10
  Triglycerides (mg/dL)
Mean Change from Post-Intervention in Insulin at 10 weeks | Post-Detraining at week 10
  Insulin (μU/mL)
Mean Change from Post-Intervention in Fasting blood glucose at 10 weeks | Post-Detraining at week 10
  Fasting blood glucose (mg/dL)
Mean Change from Post-Intervention in Body weight at 10 weeks | Post-Detraining at week 10
  Body weight (kilograms)
Mean Change from Post-Intervention in Total Body Fat Percentage at 10 weeks | Post-Detraining at week 10
  Total Body Fat Percentage (%BF): The percent of the body that is composed of fat. This will change based on the amount of fat there is as well as the amount of lean mass there is.
Mean Change from Post-Intervention in Skeletal Muscle Mass Percentage at 10 weeks | Post-Detraining at week 10
  Skeletal Muscle Mass Percentage (%SMM): The percent of the body that is composed of skeletal muscle. Like %BF, this number is relative to total mass.

SECONDARY OUTCOMES:
Mean Change from Baseline in Bacterial Profile at 4 weeks | Post-Supplementation at week 4
  Fecal Microbial DNA (16s Sequencing)
Mean Change from Baseline in Serum Acetate Profile at 4 weeks | Post-Supplementation at week 4
  Serum Acetate (SCFA: gas chromatography analysis)
Mean Change from Baseline in Fecal acetate Profile at 4 weeks | Post-Supplementation at week 4
  Fecal acetate (SCFA: in fecal samples by liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Baseline in Propionate Profile at 4 weeks | Post-Supplementation at week 4
  Propionate (liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Baseline in Butyrate Profile at 4 weeks | Post-Supplementation at week 4
  Butyrate (liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Baseline in Markers of Serum lipopolysaccharides at 4 weeks | Post-Supplementation at week 4
  Serum lipopolysaccharides (LPS, ng/ml)
Mean Change from Baseline in Markers of Serum lipopolysaccharides-binding protein at 4 weeks | Post-Supplementation at week 4
  Serum lipopolysaccharides-binding protein (LBP, pg/ml)
Mean Change from Baseline in Bacterial Profile at 8 weeks | Post-Intervention at week 8
  Fecal Microbial DNA (16s Sequencing)
Mean Change from Baseline in Serum Acetate Profile at 8 weeks | Post-Intervention at week 8
  Serum Acetate (SCFA: gas chromatography analysis)
Mean Change from Baseline in Fecal acetate Profile at 8 weeks | Post-Intervention at week 8
  Fecal acetate (SCFA: in fecal samples by liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Baseline in Propionate Profile at 8 weeks | Post-Intervention at week 8
  Propionate (liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Baseline in Butyrate Profile at 8 weeks | Post-Intervention at week 8
  Butyrate (liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Baseline in Markers of Serum lipopolysaccharides at 8 weeks | Post-Intervention at week 8
  Serum lipopolysaccharides (LPS, ng/ml)
Mean Change from Baseline in Markers of Serum lipopolysaccharides-binding protein at 8 weeks | Post-Intervention at week 8
  Serum lipopolysaccharides-binding protein (LBP, pg/ml)
Mean Change from Baseline in Serum Acetate Profile at 10 weeks | Post-Detraining at week 10
  Serum Acetate (SCFA: gas chromatography analysis)
Mean Change from Baseline in Fecal acetate Profile at 10 weeks | Post-Detraining at week 10
  Fecal acetate (SCFA: in fecal samples by liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Baseline in Bacterial Profile at 10 weeks | Post-Detraining at week 10
  Fecal Microbial DNA (16s Sequencing)
Mean Change from Baseline in Propionate Profile at 10 weeks | Post-Detraining at week 10
  Propionate (liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Baseline in Butyrate Profile at 10 weeks | Post-Detraining at week 10
  Butyrate (liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Baseline in Markers of Serum lipopolysaccharides at 10 weeks | Post-Detraining at week 10
  Serum lipopolysaccharides (LPS, ng/ml)
Mean Change from Baseline in Markers of Serum lipopolysaccharides-binding protein at 10 weeks | Post-Detraining at week 10
  Serum lipopolysaccharides-binding protein (LBP, pg/ml)
Mean Change from Post-Supplementation in Bacterial Profile at 8 weeks | Post-Intervention at week 8
  Fecal Microbial DNA (16s Sequencing)
Mean Change from Post-Supplementation in Serum Acetate Profile at 8 weeks | Post-Intervention at week 8
  Serum Acetate (SCFA: gas chromatography analysis)
Mean Change from Post-Supplementation in Fecal acetate Profile at 8 weeks | Post-Intervention at week 8
  Fecal acetate (SCFA: in fecal samples by liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Post-Supplementation in Propionate Profile at 8 weeks | Post-Intervention at week 8
  Propionate (liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Post-Supplementation in Butyrate Profile at 8 weeks | Post-Intervention at week 8
  Butyrate (liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Post-Supplementation in Markers of Serum lipopolysaccharides at 8 weeks | Post-Intervention at week 8
  Serum lipopolysaccharides (LPS, ng/ml)
Mean Change from Post-Supplementation in Markers of Serum lipopolysaccharides-binding protein at 8 weeks | Post-Intervention at week 8
  Serum lipopolysaccharides-binding protein (LBP, pg/ml)
Mean Change from Post-Intervention in Bacterial Profile at 10 weeks | Post-Detraining at week 10
  Fecal Microbial DNA (16s Sequencing)
Mean Change from Post-Intervention in Serum Acetate Profile at 10 weeks | Post-Detraining at week 10
  Serum Acetate (SCFA: gas chromatography analysis)
Mean Change from Post-Intervention in Fecal acetate Profile at 10 weeks | Post-Detraining at week 10
  Fecal acetate (SCFA: in fecal samples by liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Post-Intervention in Propionate Profile at 10 weeks | Post-Detraining at week 10
  Propionate (liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Post-Intervention in Butyrate Profile at 10 weeks | Post-Detraining at week 10
  Butyrate (liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Post-Intervention in Markers of Serum lipopolysaccharides at 10 weeks | Post-Detraining at week 10
  Serum lipopolysaccharides (LPS, ng/ml)
Mean Change from Post-Intervention in Markers of Serum lipopolysaccharides-binding protein at 10 weeks | Post-Detraining at week 10
  Serum lipopolysaccharides-binding protein (LBP, pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Kembra D Albracht-Schulte, Ph.D, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech Kinesiology Building, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No